CLINICAL TRIAL: NCT06961604
Title: A Novel Method for Determination of Thromboembolic Stroke Origin
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, jcassuto, MD, Atlantic Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2323793-1
Record Dates: First submitted 2025-05-06; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Thromboembolic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention - NaF PET (Experimental): Intervention/Experimental Arm - non-cardiogenic thromboembolic stroke patients to undergo NaF PET-CT
  Interventions: Drug: NaF PET-CT

INTERVENTIONS:
Drug: NaF PET-CT — Following a non-cardiogenic thromboembolic stroke, patients will undergo NaF PET-CT imaging to identify the culprit plaque and any other vulnerable plaques at high risk for rupture

SUMMARY:
Rupture of vulnerable carotid, vertebral, and intracranial arterial plaques results in thromboembolic stroke. Identification of these culprit lesions is an important component of post-stroke care. This study seeks to test the feasibility of NaF PET-CT to detect these plaques and alter patient care. Prior studies have shown a high degree of correlation between NaF PET+ lesions and high-risk plaque features on high resolution MRI, including mirocalcification, necrosis, and ulceration.

ELIGIBILITY:
Inclusion Criteria: 18 years of age or older with a non-cardiogenic thromboembolic stroke in the past 14 days.

Exclusion Criteria: Less than 18 years of age, any other kind of stroke, not clinically stable to undergo PET-CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Culprit lesion | Within 14 days of the stroke
  Can NaF PET-CT within 14 days of a non-cardiogenic thromboembolic stroke identify the likely culprit plaque as a source of the stroke

SECONDARY OUTCOMES:
Recurrent stroke | Within 1 year of imaging
  Can NaF PET-CT within 14 days of a non-cardiogenic thromboembolic stroke predict the location of a future non-cardiogenic thromboembolic stroke
Management change | Within 1 year of imaging
  Can NaF PET-CT within 14 days of a non-cardiogenic thromboembolic stroke alter patient management

CONTACTS AND LOCATIONS:
Locations (1):
- Overlook Medical Center, Summit, New Jersey, United States